CLINICAL TRIAL: NCT00546429
Title: Clinical Trial to Monitor the Clinical Effectiveness of the DePuy ATN Trochanteric Nailing System in the Treatment of Trochanteric Fractures of the Proximal Femur
Brief Title: DePuy Trochanteric (ATN) Nailing Clinical Outcomes Trial
Acronym: ATN
Status: Completed | Type: Observational
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 04077
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Results first posted 2010-12-10 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Femoral Fracture (Proximal)
Keywords: Proximal femoral fracture; Trochanteric fracture; Intramedullary nailing
MeSH Terms: conditions — Proximal Femoral Fractures; Hip Fractures | interventions — Fracture Fixation, Intramedullary; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Monitoring of trochanteric fractures after treatment with the ATN system.
  Interventions: Device: Intramedullary nailing

INTERVENTIONS:
Device: Intramedullary nailing — Trochanteric nailing for proximal femoral fractures.
  Other Names: Ace Trochanteric Nail (ATN) system

SUMMARY:
The purpose of this study is to monitor trochanteric fracture healing and review the performance of the ATN system.

DETAILED DESCRIPTION:
Proximal femoral fractures are among the most common femoral fractures. In the past plates and screws were often used to repair these fractures but this treatment had limitations including restricted weight bearing. Intermedullary nailing is an alternative to plate and screw treatment. Weight bearing is allowed and the procedure can be a less invasive. Among intramedullary nailing complications are iatrogenic fractures that can be further divided into trochanteric and femoral shaft fractures. Trochanteric fractures often heal without additional intervention however femoral shaft fractures usually require an additional surgical procedure to facilitate healing. This study will monitor fracture healing using clinical and radiographic evaluations of subjects with trochanteric fractures of the proximal femur treated with the ATN system.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willing to sign the approved consent form.
* 18 years of age
* Skeletally mature
* Have stable or unstable proximal femur fracture, including pertrochanteric, intertrochanteric, high subtrochanteric or any combination of the AO Proximal Femur Fracture Classification

Exclusion Criteria:

* Subjects with concomitant lower extremity injuries or multiple trauma that would interfere with normal hip fracture rehabilitation.
* Subjects who have isolated or combined medial femoral neck fractures.
* Subjects who are unwilling or unable to comply with a rehabilitation program or are unwilling or unable to be assessed for 1 year following surgery.
* Subjects who are pregnant or breastfeeding.
* Subjects who are a prisoner or a known alcohol or drug abuser.
* Subjects who have a prior surgical history in the affected hip, or conditions that may interfere with outcome or impede healing.
* Subjects who have an obliterated medullary canal or other conditions that may complicate the reaming process.
* Subjects who have evidence of active untreated infections that may spread to other areas of the body.
* Subjects who have a highly communicable disease or pathology that may limit follow-up.
* Subjects, who in the opinion of the Clinical Investigator, have an existing condition that indicates the Subject is not a good candidate for the study.
* Subjects who are participating in another clinical investigation.
* Subjects known to have allergies to titanium, aluminum, vanadium.
* Subjects who are currently eligible for workman's compensation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-09-01 (Actual); Primary Completion 2009-09-01 (Actual); Study Completion 2009-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Himden, Study Director — DePuy Orthopaedics
Locations (4):
- United States (4):
  - Front Range Orthopaedics, Colorado Springs, Colorado
  - Orthopaedic Physicians of Colorado, Englewood, Colorado
  - Erie County Medical Center, Buffalo, New York
  - Blue Ridge Bone and Joint, Asheville, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2006 & September 2009, 62 subjects were recruited and enrolled at 6 US clinics by orthopaedic surgeons. Each study site could enroll up to 20 subjects (cohorts were re-assigned as necessary to complete enrollment in a timely manner). Recruitment was based on the inclusion and exclusion criteria in the clinical investigation plan.
Pre-assignment Details: This was a non-randomized study so all subjects that met the inclusion/exclusion criteria received the ATN Trochanteric Nail. Consented subjects could be excluded from the trial based on results of pre-operative clinical and/or radiographic evaluations, as per the exclusion criteria in the clinical investigation plan.
Groups:
- DePuy Orthopaedics ATN Trochanteric Nail System: The participants in this study will undergo treatment of trochanteric fractures using DePuy Orthopaedics ATN Trochanteric Nail System implants and results will be reviewed by clinical and radiographic evaluations.
Period: Overall Study
Arm/Group | DePuy Orthopaedics ATN Trochanteric Nail System
Started | 62 (2 subjects did not have a preoperative Merle D'Aubigne score.)
Completed | 32
Not Completed | 30

BASELINE CHARACTERISTICS:
Arm/Group | DePuy Orthopaedics ATN Trochanteric Nail System
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States: United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Success in Terms of the Merle D'Aubigne Postel Score for Pain Category
Description: Merle D'Aubigne measures three categories for Pain, Mobility and Ability to walk using a 0 to 6 scoring scale for each category. Scoring is 0 indicating worse outcomes and 6 indicating better outcomes. Each Category is scored and reported separately
Time Frame: 4 weeks, 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DePuy Orthopaedics ATN Trochanteric Nail System
Number analyzed (Participants) | 60
Units on a scale
  4 Week Merle D'Aubigne for Pain Score (0 worst to 6 best) | 4.1 (1.2)
  3 Month Merle D'Aubigne Pain Score (0 worst to 6 best) | 4.4 (1.4)
  6 Month Merle D'Aubigne Pain Score (0 worst to 6 best) | 4.5 (1.3)
  12 Month Merle D'Aubigne Pain Score (0 worst to 6 best) | 4.6 (1.6)

2. Secondary Outcome: Lower Extremity Measure (LEM)
Time Frame: 4 weeks, 3, 6 and 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Medical Imaging
Time Frame: 4 weeks, 3, 6 and 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Six Item Screener and Ambulatory Status
Time Frame: 4 weeks, 3, 6 and 12 months
Reporting Status: Not Posted

5. Secondary Outcome: SF-12
Time Frame: 4 weeks, 3, 6 and 12 months
Reporting Status: Not Posted

6. Primary Outcome: Success in Terms of the Merle D'Aubigne Postel Score for Walk Category
Description: as for outcome 1
Time Frame: 4 weeks, 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DePuy Orthopaedics ATN Trochanteric Nail System
Number analyzed (Participants) | 60
Units on a scale
  4 Week Merle D'Aubigne for Walk Score (0 worst to 6 best) | 1.3 (1.3)
  3 Month Merle D'Aubigne Walk Score (0 worst to 6 best) | 2.6 (1.7)
  6 Month Merle D'Aubigne Walk Score (0 worst to 6 best) | 3.0 (1.9)
  12 Month Merle D'Aubigne Walk Score (0 worst to 6 best) | 2.7 (1.9)

7. Primary Outcome: Success in Terms of the Merle D'Aubigne Postel Score for Mobility Category
Description: as for outcome 1
Time Frame: 4 weeks, 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DePuy Orthopaedics ATN Trochanteric Nail System
Number analyzed (Participants) | 60
Units on a scale
  4 Week Merle D'Aubigne for Mobility Score (0 worst to 6 best) | 5.2 (1.3)
  3 Month Merle D'Aubigne Mobility Score (0 worst to 6 best) | 5.4 (1.0)
  6 Month Merle D'Aubigne Mobility Score (0 worst to 6 best) | 5.4 (1.0)
  12 Month Merle D'Aubigne Mobility Score (0 worst to 6 best) | 5.6 (0.8)

ADVERSE EVENTS:
Arm/Group | DePuy Orthopaedics ATN Trochanteric Nail System
Serious Adverse Events (participants affected / at risk) | 3/62
Other Adverse Events (participants affected / at risk) | 4/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DePuy Orthopaedics ATN Trochanteric Nail System (N=62)
Bone fracture acetabulum (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — This subject died and which is also noted as an adverse event in this study.
Death (General disorders) | 1 (1) — This subject suffered from cancer which is also noted as an adverse event in this study.
Implant removal (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DePuy Orthopaedics ATN Trochanteric Nail System (N=62)
Respiratory system (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less